CLINICAL TRIAL: NCT07091422
Title: A Split-Mouth Clinical Trial Evaluating the Bond Failure Rate of a New Etch-Free Orthodontic Adhesive
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Flavio Copello, Dr Flavio Copello, DDS, Principal Investigator, Clinical Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00115604
Record Dates: First submitted 2025-07-15; First posted 2025-07-29 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Bracket Bonding; Orthodontic Treatment; Dental Adhesives/Restorations Performance; White Spot Lesion of Tooth
Keywords: Etch-Free Adhesive; Orthodontic Bonding; Bracket Failure; Split-Mouth Trial; White Spot Lesions; Orthodontics Clinical Trial

STUDY DESIGN:
Intervention Model Description: Split-mouth
Who Masked: Outcomes Assessor
Masking Description: Single-blinded (Outcome Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Etch-Free Adhesive (Experimental): Teeth on one randomized side of the mouth will be bonded with a novel self-adhesive orthodontic material that does not require prior acid etching or primer application.
  Interventions: Device: Etch-Free Adhesive
- Conventional Etch-and-Bond Adhesive (Experimental): Teeth on the contralateral side of the mouth will be bonded using the standard orthodontic bonding protocol with 35-37% phosphoric acid etching, primer, and conventional resin adhesive.
  Interventions: Device: Conventional Etch-and-Bond Adhesive

INTERVENTIONS:
Device: Etch-Free Adhesive — A self-adhesive orthodontic bonding material applied directly to enamel without prior phosphoric acid etching or primer application. Brackets are bonded following the manufacturer's instructions.
  Arms: Etch-Free Adhesive
Device: Conventional Etch-and-Bond Adhesive — A standard orthodontic bonding protocol using 35-37% phosphoric acid etching, primer application, and a conventional light-cure adhesive. Brackets are bonded following the manufacturer's recommended procedure.
  Arms: Conventional Etch-and-Bond Adhesive

SUMMARY:
This randomized, split-mouth clinical trial will evaluate a new orthodontic adhesive that eliminates the need for acid etching before bracket bonding. Conventional orthodontic bonding requires etching enamel with phosphoric acid, which can weaken the outer enamel layer and increase the risk of white spot lesions and enamel damage. The etch-free adhesive under investigation is designed to simplify the bonding procedure while preserving enamel integrity.

Twenty orthodontic patients starting treatment with braces will participate. For each patient, one side of the mouth (left or right) will be randomly assigned to receive the etch-free adhesive, while the opposite side will receive the conventional adhesive with acid etching. This intra-patient design allows a direct comparison under identical oral conditions.

Participants will be followed for 12 months. Bracket failures, bonding time, ease of adhesive removal, enamel surface condition after debonding, and the presence of white spot lesions will be recorded. If effective, the etch-free adhesive may reduce enamel damage without compromising bond strength, providing a safer and more efficient bonding option for orthodontic patients.

DETAILED DESCRIPTION:
This is a prospective, randomized, split-mouth clinical trial designed to compare the bond failure rate, bonding efficiency, and enamel outcomes of a novel etch-free orthodontic adhesive with a conventional acid-etch adhesive over a 12-month follow-up period.

Background and Rationale Conventional orthodontic bonding requires phosphoric acid etching to create surface roughness for adhesive retention. While effective, this process irreversibly demineralizes enamel and may increase susceptibility to white spot lesions (WSLs), decalcification, and enamel fractures during bracket removal.

A new generation of self-adhesive bonding materials eliminates the etching step by bonding directly to enamel. This simplified approach may preserve enamel integrity, reduce chair time, and improve the patient experience while maintaining adequate bond strength.

The split-mouth design allows direct intra-patient comparison of the two bonding methods under identical oral conditions (hygiene, diet, occlusal forces), reducing inter-patient variability.

Study Design Type: Prospective, randomized, split-mouth trial

Population: 20 patients (ages ≥12 years) with permanent dentition undergoing fixed orthodontic treatment

Follow-up duration: 12 months post-bonding

Setting: University-based orthodontic clinic

Interventions Test Adhesive (Experimental): A commercially available etch-free adhesive system applied directly to enamel without acid etching or separate priming.

Control Adhesive: Conventional orthodontic adhesive applied following 37% phosphoric acid etching, primer, and adhesive placement.

Randomization and Bonding Procedure Each patient will receive both adhesives-one on the left side and one on the right-randomly assigned using a computer-generated randomization schedule and sealed envelopes.

Bonding will be performed by a calibrated operator using identical brackets and bonding techniques.

Control side: 37% phosphoric acid etch (30 seconds), rinse, dry, primer, and adhesive.

Experimental side: Etch-free adhesive applied directly per manufacturer instructions.

Bonding time for each side will be measured with a stopwatch.

Sample Size Justification Twenty patients will contribute approximately 212 bonded brackets (10-12 per side, excluding molars and second premolars). This sample size provides 80% power to detect a clinically meaningful difference in bond failure rates (expected 5% failure rate for the etch-free adhesive vs. 10% for conventional adhesive; α = 0.05), analyzed using McNemar's test for paired binary outcomes.

Outcome Measures Primary Outcome

Bracket Failure Rate: Number and location of dislodged brackets on test vs. control sides recorded at monthly visits.

Secondary Outcomes

Bonding Time: Measured in seconds per side.

Enamel Condition at Debonding: Assessed clinically and photographically by blinded evaluators.

Adhesive Remnant Index (ARI): Scored 0-3 after debonding.

White Spot Lesions (WSLs): Presence and severity assessed clinically and photographically at baseline and after 12 months using standardized scoring.

Patient-Reported Outcomes (if applicable): Discomfort related to bonding/debonding.

Data Collection and Management Data will be recorded using standardized forms and stored on secure, encrypted institutional servers.

Clinical photographs will document enamel condition and WSLs.

All data will be coded and de-identified. Only authorized study personnel will have access.

Ethical Considerations The study has been reviewed by the University of Maryland Institutional Review Board (IRB #HP-00115604) and determined to be minimal risk.

Written informed consent will be obtained from adult participants; minors will provide assent with parental consent.

Both adhesives are commercially available and widely used in clinical practice; no experimental drugs or devices are involved.

No additional radiographs or invasive procedures are required beyond standard care.

Participants may withdraw at any time without affecting their ongoing treatment.

This trial seeks to determine whether an etch-free adhesive can reduce enamel damage and improve bonding efficiency without compromising clinical performance.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 14 to 35 years

Requiring comprehensive fixed orthodontic treatment with brackets on both arches

Good general health with no contraindications to orthodontic treatment

Presence of at least 10 permanent teeth per arch suitable for bracket bonding

Ability and willingness to comply with study visits and follow-up for at least 12 months

Parent/guardian consent and child assent obtained as appropriate

Exclusion Criteria:

Presence of systemic diseases or conditions that affect oral health or healing (e.g., uncontrolled diabetes, immunosuppression)

Teeth with significant enamel defects, restorations, or caries in bonding areas

Patients currently undergoing or who have undergone orthodontic treatment previously

History of allergy or sensitivity to dental adhesives or related materials

Patients with poor oral hygiene or active periodontal disease

Use of medications known to affect tooth enamel or oral tissues (e.g., long-term corticosteroids)

Inability to attend follow-up visits or anticipated lack of compliance

Participation in another clinical trial that could interfere with study outcomes

Ages: 14 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-08-11 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Bracket Failure Rate | Through study completion, up to 12 months post-bonding (evaluated at each routine orthodontic visit).
  The proportion of brackets bonded with each adhesive (etch-free vs. conventional) that experience bond failure over a 12-month follow-up period. A bond failure is defined as a clinically detached bracket requiring rebonding.

SECONDARY OUTCOMES:
Bonding Time Per Quadrant | At the initial bonding appointment (Day 1).
  The time required to bond all brackets in one quadrant using either adhesive, measured in minutes using a digital timer.
Adhesive Remnant Index (ARI) at Debonding | At debonding (approximately 12 months post-bonding or at completion of treatment).
  The amount of adhesive remaining on the tooth surface after bracket removal, scored using the standardized Adhesive Remnant Index (0-3 scale).
Enamel Surface Integrity | At debonding (approximately 12 months post-bonding).
  Visual assessment of enamel for cracks, roughness, or damage after bracket removal, evaluated through clinical inspection and standardized digital photographs.
White Spot Lesion (WSL) Formation | At baseline (Day 1), 6 months, and 12 months post-bonding.
  Incidence and severity of new white spot lesions on bonded teeth, assessed using a standardized WSL index at 6 and 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Baltimore School of Dentistry, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
This study involves minimal-risk clinical data and will be reported in aggregate form only. De-identified individual participant data will not be shared outside the study team.